CLINICAL TRIAL: NCT02681614
Title: Pilot Study Evaluating the Role of Histopathology Correlation in Treatment Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE10814
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Imaging; Prostate; Multiparametric MRI; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Uronav (Experimental): Participants will undergo a Uronav guided biopsy with Magnetic Resonance Imaging confirmation.
  All biopsies will be completed in the outpatient setting in the ambulatory OR prior to routine prostate brachytherapy under general anesthesia.
  Interventions: Device: Uronav guided biopsy; Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Uronav guided biopsy — All biopsies will be completed in the outpatient setting in the ambulatory operating room prior to routine prostate brachytherapy under general anesthesia.
  Patients will be prepped in a dorsal lithotomy position with insertion of a Foley catheter. The perineum will be shaved as needed, and cleansed with antiseptic solution, and the scrotum will be elevated with a towel roll to expose the perineum.
  Other Names: Phillips Medical's Uronav
Device: Magnetic resonance imaging — An MRI (magnetic resonance imaging) is a scan that uses radio waves and a strong magnetic field to provide images of internal organs and tissues. This is not part of the study but will have been done per standard treatment. An MRI will occur at the screening visit and last visit of the study.
  Other Names: MRI

SUMMARY:
This clinical research study tests the Uronav system. Patients with prostate cancer will be asked to take part in this study.

Uronav system is an investigational device that is used on this study to help place markers in the patient. These are called fiducial markers and they are placed in the patient to help plan radiation treatment. Radiation therapy treatment will be planned by the treating physician and will not be experimental or part of this research study.

This study will also test the similarities and differences of biopsy tissue structures and the findings from the intraprostatic MRI (internally guided MRI).

DETAILED DESCRIPTION:
Study Objectives

Specific Aim 1: Evaluate final pathology post-operatively for histopathology confirmation of multiparametric MRI targets detected during treatment planning. This will be accomplished by using transperineal biopsies obtained prior to interstitial brachytherapy during the procedure, while under anesthetic just prior to the placement of the brachytherapy needles and sources.

Specific Aim 2: Evaluate the ability of the Uronav system in a transperineal setting to guide biopsy needle placement using the electromagnetic guidance system and transperineal ultrasound probe stabilization device and stepper.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathology confirmed prostate cancer that is Gleason score ≤7(4+3) clinical stage ≤ T2bN0M0 with a Prostate-specific antigen (PSA) below 15 ng/mL.
* Patients must have MRI findings reporting intraprostatic lesions suspicious for malignancy.
* Patient must not have had any prior treatment for prostate cancer
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Subjects must have an International Prostate Symptom Score of ≤ 15.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Gleason score of ≥ 8(4+4)
* PSA ≥ 15 ng/mL.
* Clinical stage >T2b or evidence of nodal
* Patients who are on anticoagulants or high dose aspirin therapy that cannot be safely stopped for greater than 10 days prior to treatment should be excluded to limit increased risk for urinary obstruction.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the unlikely risk of prostate cancer being life threatening in this population.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Traughber, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fredman E, Traughber B, Kharouta M, Podder T, Lo S, Ponsky L, MacLennan G, Paspulati R, Ellis B, Machtay M, Ellis R. Focal Prostate Stereotactic Body Radiation Therapy With Correlative Pathological and Radiographic-Based Treatment Planning. Front Oncol. 2021 Sep 15;11:744130. doi: 10.3389/fonc.2021.744130. eCollection 2021. PMID 34604088

RESULTS

PARTICIPANT FLOW:
Groups:
- Uronav: Participants will undergo a Uronav guided biopsy with Magnetic Resonance Imaging confirmation
  o All biopsies will be completed in the outpatient setting in the ambulatory OR prior to routine prostate brachytherapy under general anesthesia.
  Uronav guided biopsy: All biopsies will be completed in the outpatient setting in the ambulatory operating room prior to routine prostate brachytherapy under general anesthesia. Patients will be prepped in a dorsal lithotomy position with insertion of a Foley catheter. The perineum will be shaved as needed, and cleansed with antiseptic solution, and the scrotum will be elevated with a towel roll to expose the perineum.
  Magnetic resonance imaging: An MRI (magnetic resonance imaging) is a scan that uses radio waves and a strong magnetic field to provide images of internal organs and tissues. This is not part of the study but will have been done per standard treatment. An MRI will occur at the screening visit and last visit of the study.
Period: Overall Study
Arm/Group | Uronav
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Uronav
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 1
  60-69 years | 2
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Biopsies With True Positives Between Biopsy Tissue and Intraprostatic MRI
Description: Number of participants who had biopsies with true positives between biopsy tissue and intraprostatic MRI (sensitivity of the intraprostatic MRI)
Time Frame: Within 15 days of screening
Population: All participants who were put on study and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Uronav
Number analyzed (Participants) | 5
Participants | 2

2. Primary Outcome: Number of Biopsies With True Negatives Between Biopsy Tissue and Intraprostatic MRI
Description: Number of biopsies with true negatives between biopsy tissue and intraprostatic MRI (specificity of the intraprostatic MRI)
Time Frame: Within 15 days of screening
Population: All participants who were put on study and received treatment
Measure: Number; unit: biopsies
Arm/Group | Uronav
Number analyzed (Participants) | 5
biopsies | 2

3. Primary Outcome: Number of Biopsies With False Positives Between Biopsy Tissue and Intraprostatic MRI
Description: Number of biopsies with false positives between biopsy tissue and intraprostatic MRI (positive predictive values of MRI)
Time Frame: Within 15 days of screening
Population: All participants who were put on study and received treatment
Measure: Number; unit: biopsies
Arm/Group | Uronav
Number analyzed (Participants) | 5
biopsies | 1

4. Primary Outcome: Number of Biopsies With False Negatives Between Biopsy Tissue and Intraprostatic MRI
Description: Number of biopsies with false negatives between biopsy tissue and intraprostatic MRI (negative predictive values of MRI)
Time Frame: Within 15 days of screening
Population: All participants who were put on study and received treatment
Measure: Number; unit: biopsies
Arm/Group | Uronav
Number analyzed (Participants) | 5
biopsies | 2

5. Secondary Outcome: Number of Participants With Infections Within 30 Days
Description: The infection rate within 30 days due to the procedure will be collected for expected acute events and these data will be used for reporting the study results for specific aim 2 evaluation the transperineal use of Uronav to determine if the transperineal biopsy approach results in a reduced rate of infection compared to standard transrectal biopsies .
Time Frame: Up to 30 days post biopsy
Population: All participants who were put on study and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Uronav
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Number of Hospitalizations Within 30 Days
Description: The hospitalization rate within 30 days due to the procedure will be collected for expected acute events and these data will be used for reporting the study results for specific aim 2 evaluation the transperineal use of Uronav to determine if the transperineal biopsy approach results in a reduced rate of hospitalization compared to standard transrectal biopsies .
Time Frame: Up to 30 days post biopsy
Population: All participants who were put on study and received treatment
Measure: Number; unit: hospitilizations
Arm/Group | Uronav
Number analyzed (Participants) | 5
hospitilizations | 0

7. Secondary Outcome: Number of Participants Who Had Successful Completion of Transperineal Biopsy Procedure
Description: The study will be to report the incidence of successful completion of the transperineal biopsy procedure using the Uronav system which is provided by Philips Medical as part of the support for this study
Time Frame: Up to 15 days after screening
Population: All participants who were put on study and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Uronav
Number analyzed (Participants) | 5
Participants | 5

8. Secondary Outcome: Dosimetric Coverage of Brachytherapy Implant Described by Mean V100 (% Volume)
Description: Post-operative radiation dose coverage reported as volumes of prostate receiving a percentage of the prescribed dose, described by mean V100 (% volume)
Time Frame: Up to 15 days after screening
Population: All participants who were put on study and received treatment
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Uronav
Number analyzed (Participants) | 5
percent | 95.75 (0.03)

9. Secondary Outcome: Dosimetric Coverage of Brachytherapy Implant Described by Mean D90 (% Rx)
Description: Dosimetric coverage of brachytherapy implant described by mean D90 (% Rx), which refers to the main dose in the hottest 90% of the post-implant prostate volume (given as a percent of the RX dose)
Time Frame: Up to 15 days after screening
Population: All participants who were put on study and received treatment
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Uronav: Participants will undergo a Uronav guided biopsy with Magnetic Resonance Imaging confirmation.
  All biopsies will be completed in the outpatient setting in the ambulatory OR prior to routine prostate brachytherapy under general anesthesia.
  Uronav guided biopsy: All biopsies will be completed in the outpatient setting in the ambulatory operating room prior to routine prostate brachytherapy under general anesthesia.
  Patients will be prepped in a dorsal lithotomy position with insertion of a Foley catheter. The perineum will be shaved as needed, and cleansed with antiseptic solution, and the scrotum will be elevated with a towel roll to expose the perineum.
  Magnetic resonance imaging: An MRI (magnetic resonance imaging) is a scan that uses radio waves and a strong magnetic field to provide images of internal organs and tissues. This is not part of the study but will have been done per standard treatment. An MRI will occur at the screening visit and last visit of the study.
Arm/Group | Uronav
Number analyzed (Participants) | 5
percent | 111.63 (0.07)

10. Secondary Outcome: Dosimetric Coverage of Targeted Lesion Described by Mean V100 (% Volume)
Description: post-operative radiation dose coverage reported as volumes of targeted lesion receiving a percentage of the prescribed dose, described by mean V100 (% Volume)
Time Frame: Up to 15 days after screening
Population: All participants who were put on study and received treatment
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Uronav
Number analyzed (Participants) | 5
percent | 99.48 (0.01)

11. Secondary Outcome: Dosimetric Coverage of Targeted Lesion Described by Mean D90 (%Rx)
Description: Dosimetric coverage of target lesion described by mean D90 (% Rx), which refers to the main dose in the hottest 90% of the targeted lesion volume (given as a percent of the RX dose)
Time Frame: Up to 15 days after screening
Population: All participants who were put on study and received treatment
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Uronav
Number analyzed (Participants) | 5
percent | 160.83 (0.13)

ADVERSE EVENTS:
Time Frame: Patients were be followed for safety assessments at post-operative day 1, and at 2 weeks post, 1 month post, and 3 months post
Arm/Group | Uronav
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uronav (N=5)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uronav (N=5)
Nocturia (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT02681614/Prot_SAP_002.pdf
  • Informed Consent Form (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT02681614/ICF_001.pdf